CLINICAL TRIAL: NCT03502941
Title: Effect of an Essential Amino Acid/Protein Composition on Protein Metabolism
Brief Title: Effect of an EAA/Whey Composition on Protein Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 217658
Record Dates: First submitted 2018-03-30; First posted 2018-04-19 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Arm 1 and 2: Crossover design for two different doses of the product (~6.3 and 12.6 g of active components).
  Arm 3: Parallel comparison equal to the double dose of whey protein isolate (12.6 g)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A single dose of EAAs/whey (Experimental): Subjects will consume 6.3 g of EAAs/whey in ~12 oz water.
  Interventions: Dietary Supplement: 6.3 g of EAAs mixture and whey protein isolate
- A double dose of EAAs/whey (Experimental): Subjects will consume 12.6 g of EAAs/whey in ~12 oz water
  Interventions: Dietary Supplement: 12.6 g of EAAs mixture and whey protein isolate
- Whey protein alone (Experimental): Subjects will consume 12.6 g of whey protein isolate which is an equal amount to the double dose of EAAs/whey.
  Interventions: Dietary Supplement: 12.6 g of whey protein isolate

INTERVENTIONS:
Dietary Supplement: 6.3 g of EAAs mixture and whey protein isolate — A single dose of the mixture of EAAs/whey
  Other Names: Essential Blends, Fairbanks, Alaska (AK), and Pure Protein, Bayport, New York (NY)
  Arms: A single dose of EAAs/whey
Dietary Supplement: 12.6 g of EAAs mixture and whey protein isolate — A double dose of the mixture of EAAs/whey
  Other Names: Essential Blends, Fairbanks, AK, and Pure Protein, Bayport, NY
  Arms: A double dose of EAAs/whey
Dietary Supplement: 12.6 g of whey protein isolate — Whey protein isolate alone, which is an equal amount to the double dose of the mixture of EAAs/whey
  Other Names: Pure Protein, Bayport, NY
  Arms: Whey protein alone

SUMMARY:
Sarcopenia, a progressive loss of muscle mass, strength and function, is an inevitable natural process of aging. While it may be impossible to completely reverse the progress of sarcopenia, it is well established that intake of dietary protein through essential amino acids (EAAs) and whey protein increases anabolic response. The current study will test if a specially formulated mixture of EAAs and whey protein can maximally stimulate anabolic responses at the levels of whole body and muscle compared to whey protein alone.

DETAILED DESCRIPTION:
The product composition is protected by intellectual property. It contains a combination of ingredients designed to stimulate anabolic responses at whole body and muscle and to ultimately induce long-term improvements in muscle function and size. EAAs are the only dietary macronutrients that are required for survival. They are "essential" because the body cannot produce them. There are 9 dietary EAAs while there are 11 dietary non-essential amino acids that are not required in the diet because they can be produced in the body. The composition is based on a blend of 8 of the 9 EAAs. In addition to being the "active" components of dietary protein, EAAs also have the advantage over intact protein including whey protein because free EAAs are absorbed from the intestine more quickly and more completely than amino acids contained in protein, which requires digestion before absorption indicating that intact protein is relatively slowly absorbed. Therefore, the combination of free EAAs and intact protein give not only an immediate response (from the free EAAs) but also a prolonged response (from the intact protein) over time by the slower digestion. The idea of combining a specific formulation of EAAs with an intact protein to obtain both an immediate as well as a more sustained response in protein anabolism is novel. Investigators propose that consumption of the EAA/protein composition will stimulate the net protein balance at the whole body level in a dose-dependent manner. The investigators further propose that the magnitude of increase in the net protein balance will be greater than induced by the consumption of the same amount of whey protein isolate.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20 and 30 kg/m^2

Exclusion Criteria:

* Current diagnosis of diabetes
* History of malignancy in the 6 months prior to enrollment
* Weight reduction surgery
* Chronic inflammatory (Lupus, HIV/AIDS)
* Currently pregnant females
* Unable to eat dairy protein
* Unable to stop eating protein or Amino Acid (AA) supplements during the participation
* Regular resistance training (> once per week)
* Concomitant use of corticosteroids (ingestion, injection or transdermal)
* Subjects who cannot safely stop using aspirin for 7 days prior to muscle biopsies
* Hemoglobin less than 9.5 g/dL, and platelets less than 150,000 at the screening visit
* Any other disease or condition placing the subject at increased risk of harm if they were to participate, at the discretion of the study physician

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arny A Ferrando, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Park S, Church DD, Azhar G, Schutzler SE, Ferrando AA, Wolfe RR. Anabolic response to essential amino acid plus whey protein composition is greater than whey protein alone in young healthy adults. J Int Soc Sports Nutr. 2020 Feb 10;17(1):9. doi: 10.1186/s12970-020-0340-5. PMID 32041644

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 16 subjects enrolled, 8 were randomized into an arm that has a crossover component of two study interventions. The other 8 subjects were randomized into a control arm that had only one intervention.
Groups:
- EAAs/Whey (6.3 g Dose First, Then 12.6g): Subjects will consume 6.3 g of EAAs/whey in ~12 oz water at their first intervention visit, then 12.6 g of the same product at their second intervention visit.
- EAAs/Whey (12.6g First, Then 6.3g): Subjects will consume 12.6 g of EAAs/whey in ~12 oz water at their first intervention visit, then 6.3 g of the same product at their second intervention visit.
Period: Overall Study
Arm/Group | EAAs/Whey (6.3 g Dose First, Then 12.6g) | EAAs/Whey (12.6g First, Then 6.3g) | Whey Protein Alone
Started | 3 | 5 | 8
Completed | 3 | 5 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- EAAs/Whey: 6.3g First, Then 12.6g: Subjects will consume 6.3 g of EAAs/whey in ~12 oz water on 1 day. Then washout at least 5 days. Then consume 12.6 g of study product at another visit.
- EAAs/Whey: 12.6g First, Then 6.3g: Subjects will consume 12.6 g of EAAs/whey in ~12 oz water on 1 day. Then washout at least 5 days. Then consume 6.3 g of study product at another visit.
- Total: Total of all reporting groups
Arm/Group | EAAs/Whey: 6.3g First, Then 12.6g | EAAs/Whey: 12.6g First, Then 6.3g | Whey Protein Alone | Total
Number analyzed (Participants) | 3 | 5 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8 | 16
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 8
  Male | 1 | 3 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 2 | 3 | 8 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Protein Anabolism
Description: Changes in net protein balance at whole body (grams)
Time Frame: Change from 4.5 to 8.5 hours.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | A Single Dose of EAAs/Whey | A Double Dose of EAAs/Whey | Whey Protein Alone
Number analyzed (Participants) | 8 | 8 | 8
grams | 3.56 (1.89) | 11.8 (1.79) | 3.02 (0.91)
Statistical Analysis 1: Comparison: A Single Dose of EAAs/Whey vs A Double Dose of EAAs/Whey vs Whey Protein Alone; Test type: Superiority; p < 0.05, t-test, 2 sided — P value was calculated

2. Primary Outcome: Protein Synthesis
Description: Changes in protein synthesis in muscle (percent)
Time Frame: From 4.5 to 8.5 hours.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | A Single Dose of EAAs/Whey | A Double Dose of EAAs/Whey | Whey Protein Alone
Number analyzed (Participants) | 8 | 8 | 8
percent change | 0.024 (0.048) | 0.044 (0.038) | 0.022 (0.041)
Statistical Analysis 1: Comparison: A Single Dose of EAAs/Whey vs A Double Dose of EAAs/Whey vs Whey Protein Alone; Test type: Superiority; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: From enrollment to last study visit, an average of 1 month
Arm/Group | A Single Dose of EAAs/Whey | A Double Dose of EAAs/Whey | Whey Protein Alone
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT03502941/Prot_SAP_000.pdf